CLINICAL TRIAL: NCT01933490
Title: Prevention of Hypoglycemia in Patients With Post-Gastric Bypass Hyperinsulinemic Hypoglycemia
Brief Title: Post-Gastric Bypass Hypoglycemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 1306M37181
Record Dates: First submitted 2013-08-27; First posted 2013-09-02 (Estimated); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Hyperinsulinemic Hypoglycemia
Keywords: hyperinsulinemic hypoglycemia
MeSH Terms: conditions — Congenital Hyperinsulinism | interventions — Carbohydrates

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- a high carbohydrate test meal (control condition) (Other): a high carbohydrate test meal (control condition)
  Interventions: Other: high carbohydrate test meal; Other: high carbohydrate test meal after pre-treatment with rapid acting aspart insulin; Other: high fructose , low glucose test meal with carbohydrate and caloric content similar to the control meal
- high carbohydrate test meal after pre-treatment (Active Comparator): a high carbohydrate test meal after pre-treatment with rapid acting aspart insulin (insulin condition)
  Interventions: Other: high carbohydrate test meal; Other: high carbohydrate test meal after pre-treatment with rapid acting aspart insulin; Other: high fructose , low glucose test meal with carbohydrate and caloric content similar to the control meal
- high fructose low glucose test meal (Active Comparator): high fructose , low glucose test meal with carbohydrate and caloric content similar to the control meal (fructose condition)
  Interventions: Other: high carbohydrate test meal; Other: high carbohydrate test meal after pre-treatment with rapid acting aspart insulin; Other: high fructose , low glucose test meal with carbohydrate and caloric content similar to the control meal

INTERVENTIONS:
Other: high carbohydrate test meal
Other: high carbohydrate test meal after pre-treatment with rapid acting aspart insulin
Other: high fructose , low glucose test meal with carbohydrate and caloric content similar to the control meal

SUMMARY:
Post-gastric bypass hyperinsulinemic hypoglycemia is a recently described disorder occurring in some patients after gastric bypass surgery for obesity. The pathogenesis is incompletely understood but involves a robust insulin response to ingested carbohydrate. The resultant hyperinsulinemia sometimes produces hypoglycemia with neuroglycopenia, confusion and even loss of consciousness. Various treatments have been recommended including low carbohydrate diets, coingestion of the medication acarbose with carbohydrate containing meals, partial pancreatectomy and even total pancreatectomy. None is completely satisfactory. We propose to test two new potential treatments. Using a design with random assignment of three conditions we plan to compare, in 10 patients with post-gastric bypass hyperinsulinemic hypoglycemia, a high carbohydrate test meal (control condition), a high carbohydrate test meal after pre-treatment with rapid acting aspart insulin (insulin condition), and a high fructose, low glucose test meal with carbohydrate and caloric content similar to the control meal (fructose condition).

DETAILED DESCRIPTION:
Post-gastric bypass hyperinsulinemic hypoglycemia is a recently described disorder occurring in some patients after gastric bypass surgery for obesity. The pathogenesis is incompletely understood but involves a robust insulin response to ingested carbohydrate. The resultant hyperinsulinemia sometimes produces hypoglycemia with neuroglycopenia, confusion and even loss of consciousness. Various treatments have been recommended including low carbohydrate diets, coingestion of the medication acarbose with carbohydrate containing meals, partial pancreatectomy and even total pancreatectomy. None is completely satisfactory. We propose to test two new potential treatments. Using a design with random assignment of three conditions we plan to compare, in 10 patients with post-gastric bypass hyperinsulinemic hypoglycemia, a high carbohydrate test meal (control condition), a high carbohydrate test meal after pre-treatment with rapid acting aspart insulin (insulin condition), and a high fructose, low glucose test meal with carbohydrate and caloric content similar to the control meal (fructose condition). The hypothesis to be tested are 1) pretreatment with aspart insulin will prevent, or at least reduce, the occurrence of hypoglycemia and 2) substitution of fructose for glucose in the test meal will prevent, or at least reduce, the occurrence of hypoglycemia. Plasma glucose and serum insulin will be sampled before and for four hours after the three test conditions. The primary study endpoint will be the occurrence or not of plasma glucose < 60 mg/dL after the test meals. The control meal will be compared to the insulin pre-treated test meal and, in a separate comparison, to the fructose test meal. Secondary endpoints will be comparisons between the control and active treatments in peak postprandial serum insulin, peak postprandial plasma glucose, nadir postprandial plasma glucose, and the 4-hr longitudinal course of plasma glucose measurements.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be at least 21 years of age
* History of postprandial hypoglycemia with neuroglycopenia occurring one year or more after gastric bypass surgery
* History of spontaneous correction of hypoglycemia
* Normal fasting plasma glucose and serum insulin after a carbohydrate containing mixed meal, demonstration of serum insulin > 50u/UL and plasma glucose < 50mg/dL

Exclusion Criteria:

* Under 21 years of age

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-08; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
The primary study endpoint will be occurrence or not of plasma glucose < 60 mg/dL during the 4 hours after the test meal (binary endpoint). | 4 hours after meal
  The primary study endpoint will be occurrence or not of plasma glucose < 60 mg/dL during the 4 hours after the test meal (binary endpoint).

CONTACTS AND LOCATIONS:
Overall Officials: John Bantle, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Bantle AE, Wang Q, Bantle JP. Post-Gastric Bypass Hyperinsulinemic Hypoglycemia: Fructose is a Carbohydrate Which Can Be Safely Consumed. J Clin Endocrinol Metab. 2015 Aug;100(8):3097-102. doi: 10.1210/jc.2015-1283. Epub 2015 Jun 2. PMID 26037514